CLINICAL TRIAL: NCT04820140
Title: Assessment of Professional Practices in Muscle Rehabilitation of Chronic Hemodialysis
Acronym: REHABIMUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0031
Record Dates: First submitted 2021-03-19; First posted 2021-03-29 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease patient on dialysis (stage 5D); Muscle mass and strength; Training; Survival
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- muscle strengthening program: All patients will be receiving a muscle strengthening program consisting in both a training against resistance and an endurance training by elliptical bike during an observational period of 12 weeks for each treatment. Each training program will be preceded by a 4-week period of lymphatic drainage in order to improve neuromuscular sensitivity.
  Interventions: Procedure: Lymphatic drainage

INTERVENTIONS:
Procedure: Lymphatic drainage — Lymphatic drainage

SUMMARY:
Aim of this study is to evaluate, in a population of chronic kidney disease patients on dialysis (Stage 5D), the effect of a muscle strengthening program (training against resistance vs endurance training by elliptical bike) during a observational period (12 weeks per program) on frailty, risk of falling, muscle strength and mass, endurance, physical activity, quality of dialysis, nutritional status and neuromuscular sensitivity.

ELIGIBILITY:
Inclusion criteria:

* Chronic Kidney Disease patient on dialysis (stage 5D) for more than 3 months
* Age > 18 years old
* Stable clinical condition
* Absence of musculoskeletal disorders

Exclusion criteria:

* Cardiovascular contraindication
* Amputation of lower limb not allowing use of elliptical bike

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients issued from dialysis units (clinic)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Change in functional autonomy (frailty) after training | 4 weeks after inclusion
  Change in functional autonomy (frailty) after training
Change in functional autonomy (frailty) after training | 12 weeks after inclusion
  Change in functional autonomy (frailty) after training
Change in functional autonomy (frailty) after training | 16 weeks after inclusion
  Change in functional autonomy (frailty) after training and endurance training by elliptical bike during an observational period (12 weeks per program).
Change in functional autonomy (frailty) after training | 32 weeks after inclusion
  Change in functional autonomy (frailty) after training and endurance training by elliptical bike during an observational period (12 weeks per program).

SECONDARY OUTCOMES:
Change in risk of falling after training | 4, 12, 16 and 32 weeks after inclusion
  Change in risk of falling after training
Change in muscle strength and mass after training | 4, 12, 16 and 32 weeks after inclusion
  Change in muscle strength and mass after training
Change in endurance after training | 4, 12, 16 and 32 weeks after inclusion
  Change in endurance after training
Change in physical activity after training | 4, 12, 16 and 32 weeks after inclusion
  Change in physical activity after training
Change in quality of dialysis after training | 4, 12, 16 and 32 weeks after inclusion
  Change in quality of dialysis after training
Change in nutritional status after training | 4, 12, 16 and 32 weeks after inclusion
  Change in nutritional status after training
Change in neuromuscular sensitivity after training | 4, 12, 16 and 32 weeks after inclusion
  Change in neuromuscular sensitivity after training

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, Prof, Study Director — CHU Lapeyronie, Department of Biochemistry and Hormonology, Montpellier, FRANCE
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC